CLINICAL TRIAL: NCT02366520
Title: Using a Handheld Mirror to Improve Child's Behavior During Dental Treatment
Brief Title: Handheld Mirror to Improve Child's Behavior During Dental Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Masahiro Heima, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 03-14-37
Record Dates: First submitted 2015-02-09; First posted 2015-02-19 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Behavior
Keywords: Child; Child Behavior; Dental Anxiety/prevention & control; Dental Anxiety/psychology; Cooperative Behavior; Dental Care/psychology*; Humans; Videotape Recording
MeSH Terms: conditions — Behavior; Child Behavior; Cooperative Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control visit (No Intervention): The child receives dental treatment without the handheld mirror. The child cannot see the dental treatments that are conducted in his or her mouth.
- intervention visit (Experimental): The child receives dental treatment with handheld mirror. The child may see the dental treatments that are conducted in his or her mouth by the handheld mirror.
  Interventions: Device: handheld mirror

INTERVENTIONS:
Device: handheld mirror — The child may see the dental treatments that are conducted in his or her mouth by a handheld mirror.
  Arms: intervention visit

SUMMARY:
The purpose of this study is to determine whether a handheld mirror helps to reduce child behavior problems during dental treatment. It will be tested by randomized crossover design. Child participants will receive dental treatment under two conditions: during one of the treatment days the child will be given a handheld mirror; another treatment will be done without the child having the mirror. Each condition will be assign on separate days, and the day, which the child has the mirror, will be assigned by chance.

DETAILED DESCRIPTION:
Participants, including 3-17 years old children and primary caregivers as well as pediatric dentists and dental assistants, will be recruited at the Irving and Jeanne Tapper Pediatric Dental Center at University Hospitals Rainbow Babies & Children's Hospital in Cleveland, Ohio. Instructional sessions will provide proper use of a handheld mirror to pediatric dentists and dental assistants.

On the first dental appointment:

After obtain consent and assent form, the caregiver will be asked to complete a questionnaire, "Questionnaire for Caregiver", which includes questions to assess the caregiver's dental anxiety level, the caregiver's perception of the child's dental fear level, and collect characteristic information such as age and gender. The child will also be asked to complete a questionnaire; a 3-6 years old child will complete the questionnaire "Questionnaire for Child 3-6," which includes the face image scale to measure his/her level of dental anxiety; a 7-17 years old child will complete the questionnaire "Questionnaire for Child 7-17," which includes the face image scale and the Dental Subscale of the Children's Fear Survey Schedule (CFSS-DS) to measure his/her level of dental anxiety.

The child will then be randomly assigned to either Group 1, in which the child will receive the dental treatment with the mirror at the first visit and receive dental treatment without the mirror at the second visit, or Group 2, which will receive dental treatment without the mirror on the first visit and receive dental treatment with the mirror on the second visit. The child's, dentists' and dental assistants' behavior will be video recorded during treatment. The dentist will guide the child to see the inside of his or her mouth during the dental care procedure. At the end of appointment, children who are 7 -17 years old will be asked the ease of receiving dental treatment by a 5 point Likert scale.

On the second appointment, the same procedure will occur including the questionnaire and video recording.

However, the child who has been assigned to Group 1 will not have a mirror and the child who has been assigned to Group 2 will have a mirror during dental procedures.

The questionnaire and video files will be stored in a secure location which protected passwords.

Behavioral data will be coded, counted and assessed.

The child's chart will be reviewed to find the child's temperament and to count the total number of primary teeth, permanent teeth, decayed, filled, and extracted teeth due to dental caries at the examination visit.

Data analyses:

The impact of the mirror will be measured by the following variables and analyzed using the children's behavior after controlling for the children's characteristic and procedures:

1. Subject characteristic analysis
2. Comparison of variables of behavior between study group and control group after controlling for the subject's characteristics and dental treatment procedures

ELIGIBILITY:
Inclusion Criteria:

* A dyad of children who are 3-17 years of age and their primary caregiver
* Children who need at least two restorative appointments
* Primary caregivers who are fluent in English

Exclusion Criteria:

* Children who have a visual impairment
* Children who need protective stabilization to immobilize children's body for treatment
* Children who are not able to hold the mirror
* Children who don't have ability to answer the questions

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2015-05; Primary Completion 2021-04 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Number of instances of child's disruptive behavior defined by the Anxious and Disruptive Behavior Code | Child's disrupted behavior will be measured for the duration of dental treatment (up to 1 hour).
  The Anxious and Disruptive Behavior Code which includes head movement, body movement, complaints and crying, and restraints is used to count child's disrupted behavior during dental treatment.

SECONDARY OUTCOMES:
Child's cooperative behavior level assessed by Frankle's Cooperative Behavior Scale | Child's cooperative behavior will be measured for the duration of dental treatment (up to 1 hour).
  Frankle's cooperative behavior scale (Definitely negative, Negative, Positive, and Definitely positive) is used to assess child's cooperative behavior during dental treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Heima, DDS, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals, Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thrash WJ, Russel-Duggan J, Mizes JS. The origin and prevention of dental fears. Clin Prev Dent. 1984 Sep-Oct;6(5):28-32. No abstract available. PMID 6333311
- [Background] Armfield JM, Heaton LJ. Management of fear and anxiety in the dental clinic: a review. Aust Dent J. 2013 Dec;58(4):390-407; quiz 531. doi: 10.1111/adj.12118. PMID 24320894
- [Background] Milgrom P, Weinstein P, Heaton LJ. Treating fearful dental patients: a patient management handbook. 3rd edn. Seattle, WA: Dental Behavioral Resources, 2009.
- [Background] Piaget, J: The psychology of the child. New York: Basic Books, 1972
- [Background] Bandura A: Self-efficacy. San Diego, CA, Academic Press, 1994.
- [Background] Glanz K, Rimer BK, Viswanath K: Health behavior and health education: Theory, research, and practice in. San Francisco, John Wiley & Sons, Inc, 2008, p 552 p.